CLINICAL TRIAL: NCT00625768
Title: A Phase I Study of AS1409 in Patients With Either Metastatic Renal Cell Carcinoma or Metastatic Malignant Melanoma
Brief Title: Study of AS1409 in Patients With Either Metastatic Renal Cell Carcinoma or Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antisoma Research (Industry)
Responsible Party: Chris Elston, Communications Manager, Antisoma Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS1409-101
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Metastatic Renal Cell Carcinoma; Metastatic Malignant Melanoma
Keywords: Antibody; safety; tolerability; efficacy; metastatic renal cell carcinoma; metastatic malignant melanoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Melanoma | interventions — AS1409 protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: AS1409 — Study drug
  Other Names: huBC1-huIL-12

SUMMARY:
To determine the tolerability, safety, end-organ toxicity and maximum tolerated dose of AS1409 in single and repeated doses.

DETAILED DESCRIPTION:
* To determine the tolerability, safety, end-organ toxicity and maximum tolerated dose (MTD) of AS1409 in single and repeated doses.
* To determine biological responses to AS1409, including interferon-γ and IP-10 circulating concentrations.
* To determine preliminary pharmacokinetics of AS1409.
* To determine the immunogenicity of AS1409
* To explore the anti-tumour activity of AS1409.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older at the time of giving informed consent.
* Histologically confirmed diagnosis of renal cell carcinoma or malignant melanoma.
* If renal cell carcinoma, of clear cell or chromophilic/papillary type, with metastases at any site (but excluding patients with single bony lesion only).
* If malignant melanoma, unresectable Stage III disease or Stage IV disease, with metastases at any site (but excluding patients with single bony lesion only)
* Patients with clinically stable CNS metastases may enter who have been treated with surgery or radiation and who do not require steroid therapy.
* ECOG performance status 0-2.
* Patients who have received prior systemic treatment for their malignancy with chemotherapeutic or biological therapies may enter, provided treatment was completed within 4 weeks of study entry.
* Patients who have received prior experimental therapy may enter, provided treatment was completed within 12 weeks of study entry.
* Have adequate bone marrow function as evidenced by neutrophils >1.5 x109/L and platelets >100 x109/L.
* Have adequate liver and kidney function, as shown by serum bilirubin ≤1.5x upper limit of normal for the laboratory; ALT and AST both ≤2x upper limit of normal; and creatinine ≤1.5x upper limit of normal.
* Have either evaluable or measurable disease (patients entering an ascending dosage cohort) or measurable disease (patients entering the study after MTD is defined).
* Patients who have failed and or are ineligible for standard first line therapy (in accordance with individual institutional practice)

Exclusion Criteria:

Patients with any of the following will be excluded from the study:

* Patients at poor medical risk because of non-malignant systemic disease or active infection.
* History of clinically significant autoimmune or predominantly Th1-driven clinical disorders (such as rheumatoid arthritis, psoriasis, chronic inflammatory bowel disease, for example), with the exception of autoimmune endocrinopathies now treated with replacement therapy.
* Diabetic retinopathy.
* Substantive surgery within 4 weeks prior to study entry, or expectation of surgery during the study period.
* Malignancy other than renal cell carcinoma or malignant melanoma within 5 years of study entry, except for non-melanoma skin cancer and cervical intraepithelial neoplasia treated definitively or other cancer from which the patient has been disease-free for 5 years.
* Concurrent treatment with systemic steroids or with other immunosuppressive therapies.
* If female, pregnant or breastfeeding;
* Women of child bearing potential or sexually active males, unless (1) the patient (if female, or the patient's partner, if male) is surgically sterile or (2) using adequate contraception (defined as either IUD, oral or depot contraceptive, or barrier plus spermicide) while receiving study treatment and for at least 6 months after termination of treatment. Women must be post-menopausal for at least 2 years to be considered of non-childbearing potential
* Any concurrent medical or psychological condition that would limit the ability of the patient to provide informed consent or to comply with the obligations of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Tumor assessment | 6 weeks, response confirmed at 4 weeks
Biomarkers (interferon-γ and IP-10 Interferon) | Various timepoints cycles 1-6, pre- and post-dose; then 1,4 and 12 weeks post last dose
Adverse event monitoring | Various timepoints cycles 1-6, pre- and post-dose; then 1,4 and 12 weeks post last dose

CONTACTS AND LOCATIONS:
Overall Officials: James Spicer, MD, Principal Investigator — Kings College School of Medicine
Locations (4):
- New Zealand (2):
  - Auckland Medical School, Auckland
  - Waikato DHB, Hamilton
- United Kingdom (2):
  - Guys Hospital, London
  - Charing Cross Hospital, London

REFERENCES:
- [Derived] Rudman SM, Jameson MB, McKeage MJ, Savage P, Jodrell DI, Harries M, Acton G, Erlandsson F, Spicer JF. A phase 1 study of AS1409, a novel antibody-cytokine fusion protein, in patients with malignant melanoma or renal cell carcinoma. Clin Cancer Res. 2011 Apr 1;17(7):1998-2005. doi: 10.1158/1078-0432.CCR-10-2490. Epub 2011 Mar 29. PMID 21447719
- See also: Click here for additional information of Antisoma, the company sponsoring this study — http://www.antisoma.com